CLINICAL TRIAL: NCT00917410
Title: Assessment of the Health Related Effects of Compliance Optimization in Asthma Through Use of SMS (Short Message System) - A Controlled Trial
Brief Title: Mobile Phone Text for Optimizing Asthma Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: MedicoMonitor Aps (Unknown); The Ministry of Health and Prevention, Denmark (Other Government)
Responsible Party: Claus Møldrup, Associate Professor PhD, University of Copenhagen
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UC-SMS-01
Record Dates: First submitted 2009-06-05; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SMS intervention (Experimental)
  Interventions: Behavioral: SMS support

INTERVENTIONS:
Behavioral: SMS support — The intervention consisted of sequences of SMS messages sent to the intervention group, each containing 2 or 3 monitoring questions and one reminder to take the preventive medication. The SMS sequence was as follows.
  1. Remember to take your preventive asthma medication (sent at 8.00 am).
  2. Were you awakened during the night due to your asthma? Answer YES or NO.
  3. How many times have you taken your asthma attack medication during the last 24 hours? Answer a number.
  4. What was your peak flow this morning? Answer a number (optional, depending on the participant's use of a spirometer prior to the study).

SUMMARY:
The study aims at providing information on how the Short Message Service (SMS) tool influences self-management in asthma patients and to assess the resulting health related effect. A wide range of models and theories exist in the compliance area, such as technical models, communication models, cognitive models and self-management models and theories. The use of some of these theories and models will serve as theoretical and explanatory tools for studying how and why the SMS tool influences the patient's self-management.

Objective:

The objective of this study is to assess the health-related effects of a SMS compliance and monitoring system for optimized asthma treatment in a controlled trial setting.

ELIGIBILITY:
Inclusion Criteria:

* asthmatics

Exclusion Criteria:

* below 18 and above 45
* COPD patients
* no mobile phone
* not using the prescribed asthma inhalation medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Asthma control test
EQ-5D | 0, 45, 90 days
Use of health services | 0, 45, 90 days
Use of preventive medicine | 0, 45, 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Claus Møldrup, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark